CLINICAL TRIAL: NCT06498024
Title: Assessing the Blood Glucose Response of Novel Wild Rice Enhanced Food Products (ABWE) Study
Brief Title: Blood Glucose Response of Novel Wild Rice Enhanced Food Products (Trial 2)
Acronym: ABWE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The wild rice cereal development was stopped, so the trial was also withdrawn prior to starting.
Sponsor: Dylan MacKay (Other)
Collaborators: Mitacs (Industry)
Responsible Party: Sponsor-Investigator, Dylan MacKay, Assistant Professor, University of Manitoba
Organization: University of Manitoba (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HS25756 (B2022:104) (Trial 2)
Record Dates: First submitted 2024-07-04; First posted 2024-07-12 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Blood Glucose
Keywords: glycemic response; glycemic control; rice; cereal
MeSH Terms: interventions — Milk

STUDY DESIGN:
Intervention Model Description: The project will consist of 2 acute double-blind cross-over trials. The trials will follow the same study design but investigate 2 types of wild rice products. The wild rice products will be provided by the Myera group.
Who Masked: Participant, Investigator
Masking Description: The allocation of this intervention order will be blinded for the investigators and the participants. Treatment will be given blinded names, such as A and B, but it may be possible to determine what each treatment is due to its appearance, however we will not be informing the participants what the treatments are. The study staff who will be preparing and overseeing the treatments may not be blinded due to the different appearances of the treatments. However, the staff that will conduct the trial results analyses will not be un-blinded until the analyses are complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Consumption of 1 of 2 control rice cereal products (Active Comparator): This arm will provide one of the 2 white rice control products and there will be a minimum of three days separating each visit.
  Interventions: Other: Kellogg's - rice krispies (control)
- Final consumption of 1 of 2 control rice cereal products (Active Comparator): This arm will provide one of the 2 white rice control products and there will be a minimum of three days separating each visit.
  Interventions: Other: Kellogg's - rice krispies (control) + 125ml milk
- Consumption of 1 of 4 rice products (Experimental): This arm will provide 1 of the 4 randomly assigned rice products to the participant and there will be a minimum of three days separating each visit.
  Interventions: Other: Novel cereal (40% Canadian wild rice, 60% fava bean blend) + 125 ml milk
- Second consumption of 1 of 4 rice products (Experimental): This arm will provide 1 of the 4 randomly assigned rice products to the participant and there will be a minimum of three days separating each visit.
  Interventions: Other: Novel cereal (40% Canadian wild rice, 60% fava bean blend)
- Third consumption of 1 of 4 rice products (Experimental): This arm will provide 1 of the 4 randomly assigned rice products to the participant and there will be a minimum of three days separating each visit.
  Interventions: Other: Novel cereal (40% Canadian wild rice, 50% fava bean blend) + 10% purple powder (sweet potato)
- Final consumption of 1 of 4 rice products (Experimental): This arm will provide 1 of the 4 randomly assigned rice products to the participant.
  Interventions: Other: Novel cereal (40% Canadian wild rice, 50% fava bean blend) + 10% purple powder (sweet potato) + 125 ml milk

INTERVENTIONS:
Other: Kellogg's - rice krispies (control) — One serving size (140g) of whole white rice cereal will be provided. Preparation will be consistently maintained throughout.
  Arms: Consumption of 1 of 2 control rice cereal products
Other: Kellogg's - rice krispies (control) + 125ml milk — One serving size (140g) of whole white rice cereal with 125ml of milk will be provided. Preparation will be consistently maintained throughout.
  Arms: Final consumption of 1 of 2 control rice cereal products
Other: Novel cereal (40% Canadian wild rice, 60% fava bean blend) + 125 ml milk — One serving size (140g) of novel cereal (40% Canadian wild rice, 60% fava bean blend) with 125ml of milk will be provided. Preparation will be consistently maintained throughout.
  Arms: Consumption of 1 of 4 rice products
Other: Novel cereal (40% Canadian wild rice, 60% fava bean blend) — One serving size (140g) of novel cereal (40% Canadian wild rice, 60% fava bean blend) will be provided. Preparation will be consistently maintained throughout.
  Arms: Second consumption of 1 of 4 rice products
Other: Novel cereal (40% Canadian wild rice, 50% fava bean blend) + 10% purple powder (sweet potato) — One serving size (140g) of novel cereal (40% Canadian wild rice, 60% fava bean blend) with a 10% added purple powder (sweet potato) will be provided. Preparation will be consistently maintained throughout.
  Arms: Third consumption of 1 of 4 rice products
Other: Novel cereal (40% Canadian wild rice, 50% fava bean blend) + 10% purple powder (sweet potato) + 125 ml milk — One serving size (140g) of novel cereal (40% Canadian wild rice, 50% fava bean blend) and 10% purple powder (sweet potato) with 125 ml milk. Preparation will be consistently maintained throughout.
  Arms: Final consumption of 1 of 4 rice products

SUMMARY:
The goal of this acute double-blind cross over trial to test the effects of different wild rice cereal products compared to products currently on the market on glycaemic control. The main questions it aims to answer are:

1. What is the effect compared to products currently on the market on glycaemic control?
2. Is the wild rice product palatable?

Participants will:

* consent to attend 6 study visits being 2.5 hours each
* come to each visit fasted for at least 10-12 hours.
* complete a Motivation to Eat VAS following each blood measure

DETAILED DESCRIPTION:
The study will consist of 2 acute double-blind cross-over trials and both trials investigate types of wild rice products tested against a white rice or white bread control. This is the second of the two trials and will be assessing four wild rice cereals against two control rice cereals.

Participants will fast and arrive at the RCFTR between 8 and 10:30 am on the session day. They will be provided either of the study treatment based on randomization sequence. Baseline blood glucose (0 min) will be measured twice via finger stick blood sample right before their first bite of the study product, and at 15, 30, 45, 60, 90 and 120 mins after baseline in duplicate. The timer will be started when they take their first bite. VAS will be completed following consumption of the treatments to measure palatability.

The primary objective is to test the effects of different wild rice products compared to products currently on the market by evaluating factors that influence glycemic response to wild rice in humans, performed via the finger stick blood glucose that will be measured throughout each session as outlined above.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial
* Male or female between 18-50 years old
* BMI range in between 18.9-29.9 kg/m2
* Fasting glucose <5.6 mmol/L
* Usually eat breakfast
* Participant must receive at least two doses of COVID-19 vaccine that have been recognized by Winnipeg Regional Health Authorities.
* In the Investigator's opinion is able and willing to comply with all trial requirements

Exclusion Criteria:

* Fasting glucose ≥ 5.6 mmol/L or <3.5 mmol/L
* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial
* Participants who indicate that they could not finish study treatments within 10 minutes
* Use of medication or supplements that may influence carbohydrate metabolism, including, not limit to adrenergic blockers, diuretics, thiazolidinediones, metformin and systemic corticosteroids within 4 weeks of screening visit
* History of disordered eating, AIDS, hepatitis, a history of clinically important endocrine (including Type I and Type II diabetes mellitus), cardiovascular (including but not limit to atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), pulmonary, biliary or GI disorders
* Intolerance or allergic reaction to rice
* Existing restrictive dietary habits (such a vegan, low carbohydrate/keto) Date and version No: December 12 , 2022, Version 2 Page 7 of 15
* History of hypertension
* History of cancer within the last two years (except for non-melanoma skin cancer)
* Recent history (within 12 month of screening) or current consumption of >14 drinks per week, (1 drink = 12oz of beer, 5oz of wine or 1.5oz distilled spirits)
* Body weight change over 3.5kg for the past 3 months
* Participants who have participated in another research trial involving an investigational product in the past 12 weeks
* Had significant physical trauma or major surgery in the past 3 month or had trauma or major surgery in the past 3 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
The effects of different wild rice products compared to products currently on the market on glycaemic control. | Capillary blood glucose will be measured at 0 (baseline) and then 15, 30, 45, 60, 90 and 120 mins after the first bite of treatment.
  Finger stick blood glucose will be measured throughout each session.

SECONDARY OUTCOMES:
To measure the palatability of the wild rice products following consumption. | VAS measuring palatability will be completed right after the consumption of the treatments.
  Visual Analogue Scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Dylan MacKay, PHD, Principal Investigator — University of Manitoba
Locations (1):
- Chronic Disease Innovation Centre, Seven Oaks Hospital, Winnipeg, Manitoba, Canada